CLINICAL TRIAL: NCT07294677
Title: CApivasertib, Venetoclax And Low-intensity chemotheRapY for Adults With ALL/LBL
Brief Title: Trial to Test Safety of Adding Capivasertib to a Standard Leukemia Treatment Regimen
Acronym: CAVALRY
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-1773
Record Dates: First submitted 2025-12-12; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Leukemia; Lymphoma
Keywords: Chemotherapy
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — capivasertib; venetoclax; Rituximab; blinatumomab; nelarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 - Dose Escalation (Dose Level 1) (Experimental): In this arm, a dose of 320 mg dose of capivasertib will be tested in combination with venetoclax and mini-hyperCVD chemotherapy regimen.
  Interventions: Drug: Capivasertib; Drug: Venetoclax; Drug: Rituximab; Drug: Blinatumomab; Drug: Nelarabine; Drug: mini-hyperCVD
- Cohort 1 - Dose Escalation (Dose Level 2) (Experimental): In this arm, a dose of 400 mg dose of capivasertib will be tested in combination with venetoclax and mini-hyperCVD chemotherapy regimen.
  Interventions: Drug: Capivasertib; Drug: Venetoclax; Drug: Rituximab; Drug: Blinatumomab; Drug: Nelarabine; Drug: mini-hyperCVD
- Cohort 1 - Dose Escalation (Dose Level -1) (Experimental): In this arm, a dose of 200 mg dose of capivasertib will be tested in combination with venetoclax and mini-hyperCVD chemotherapy regimen.
  Interventions: Drug: Capivasertib; Drug: Venetoclax; Drug: Rituximab; Drug: Blinatumomab; Drug: Nelarabine; Drug: mini-hyperCVD
- Cohort 2 (Expansion) (Experimental): In this arm, the best, safe dose of capivasertib found after completion of enrollment to dose escalation (cohort 1) arms, will be tested in combination with venetoclax and mini-hyperCVD chemotherapy regimen.
  Interventions: Drug: Capivasertib; Drug: Venetoclax; Drug: Rituximab; Drug: Blinatumomab; Drug: Nelarabine; Drug: mini-hyperCVD
- Cohort 3 -- Arm 1 -- mini-hyperCVD + venetoclax (Randomized) (Active Comparator): Participants randomized to this arm will receive mini-hyperCVD + venetoclax.
  Interventions: Drug: Venetoclax; Drug: Rituximab; Drug: Blinatumomab; Drug: Nelarabine; Drug: mini-hyperCVD
- Cohort 3 -- Arm 2 -- mini-hyperCVD + venetoclax + capivasertib (Randomized) (Experimental): Participants randomized to this arm will receive mini-hyperCVD + venetoclax and capivasertib.
  Interventions: Drug: Capivasertib; Drug: Venetoclax; Drug: Rituximab; Drug: Blinatumomab; Drug: Nelarabine; Drug: mini-hyperCVD

INTERVENTIONS:
Drug: Capivasertib — Capivasertib taken by mouth, twice daily. Dosing will occur on a 4 days on, 3 day off schedule.
  Other Names: TRUQAP
  Arms: Cohort 1 - Dose Escalation (Dose Level -1); Cohort 1 - Dose Escalation (Dose Level 1); Cohort 1 - Dose Escalation (Dose Level 2); Cohort 2 (Expansion); Cohort 3 -- Arm 2 -- mini-hyperCVD + venetoclax + capivasertib (Randomized)
Drug: Venetoclax — Venetoclax will be taken by mouth, once daily.
  Other Names: VENCLEXTA
Drug: Rituximab — Some participants will receive rituximab by IV infusion, two doses per cycle during the first four cycles. Whether or not this will be given to participants with leukemia cells that express a protein called CD20.
  Other Names: RITUXAN
Drug: Blinatumomab — Some participants will receive cycles of blinatumomab by IV continuous infusion after the initial venetoclax plus chemotherapy phase for a 42-day cycle. Each cycle includes 28 days of blinatumomab dosing followed by a 14-day rest period. This will be given to participants that have a certain type of leukemia call CD19+ B-lineage ALL and who experience a complete remission.
  Other Names: BLINCYTO
Drug: Nelarabine — Some participants in Cohorts 1 and 2 will receive nelarabine after cycles 2 and 4 at the discretion of their treating physician.
  Other Names: ARRANON
Drug: mini-hyperCVD — Participants will receive 8 cycles of chemotherapy consisting of the following drugs.
  They will receive the part A regimen and part B regimen in alternating cycles.
  Part A: cyclophosphamide, vincristine, dexamethasone
  Part B: high dose methotrexate and cytarabine.

SUMMARY:
This is a 3-part study to assess the safety of adding capivasertib to a standard of care treatment regimen consisting of venetoclax and low-intensity chemotherapy. This chemotherapy regimen called mini-hyperCVD consists of the chemotherapy drugs, cyclophosphamide, vincristine, dexamethasone; (part A) alternating with high-dose methotrexate and cytarabine (part B) administered approximately every 28 days.

In the first part of the study (Cohort 1), the study seeks to determine the recommended dose of capivasertib that can be safely given with venetoclax and chemotherapy. Several doses of capivasertib may be tested in small groups of subjects in this part of the study. The dose tested will be increased or lowered depending on types and frequency of side effects seen until the best, safe dose is found.

Once the recommended, safe dose of capivasertib is found, the study will move on to the second part (Cohort 2) and will treat additional participants to learn more about the safety of giving these drugs together.

If the combination is determined to be safe overall, the study will move on to the third part (Cohort 3). In this part of the study, participants will be randomized to receive the mini-hyperCVD and venetoclax alone or with capivasertib.

ELIGIBILITY:
COHORT 1 Inclusion Criteria

* Patients with acute leukemia with lymphoid lineage (B-ALL, T-ALL, ETP-ALL, mixed phenotype or bi-phenotypic) or lymphoblastic lymphoma (B- or T-lineage) that is relapsed or refractory

  * Bone marrow or peripheral blood involvement with ≥5% leukemic blasts. Patients with isolated extramedullary disease that is measurable by CT scan are also eligible.
* 18 years or older
* ECOG performance status 0-2
* Adequate organ function meeting protocol criteria
* Patients must be at least 2 weeks from major surgery or radiation therapy. A wash-out period of 5 half-lives is required for patients who participated in other investigational trials. These patients must have recovered from clinically significant toxicities related to these prior treatments.
* Patients must voluntarily sign and date an informed consent prior to the initiation of any screening or study-specific procedures.
* Females of childbearing potential will use effective contraception during protocol treatment and for at least 8 months after the last dose. Males with female partners of reproductive potential will use effective contraception during protocol treatment and for at least 5 months after the last dose.

Exclusion criteria

* Ph-positive ALL, Burkitt's leukemia/lymphoma
* Patient is pregnant or breastfeeding
* Patients with uncontrolled infection.
* Known active hepatitis B or C infection, or uncontrolled human immunodeficiency virus (HIV) infection. Patients with HIV infection, whose disease is controlled with anti-retroviral therapy are eligible, but their highly active antiretroviral therapy (HAART) should be modified to minimize drug interactions. Due to the increased risk of hepatitis B reactivation, all patients with active, previously treated or resolved hepatitis B infection will not be eligible for rituximab treatment if their leukemia expresses >1% CD20.
* Major surgery or radiation therapy within 2 weeks prior to the first study dose
* Symptomatic central nervous system (CNS) disease or spinal cord compression
* Concurrent active malignancy requiring treatment with potential to influence the endpoint of the clinical trial. Patients with non-melanoma skin cancer, carcinoma in situ of the cervix, localized prostate cancer, past history of malignancy that has been definitively treated, and patients treated with hormonal therapies for solid tumors are eligible. Patients with history of multiple myeloma that does not need active treatment are also eligible.
* Uncontrolled cardiac disease
* Uncontrolled diabetes mellitus, defined as fasting blood glucose >160 mg/dL or random blood glucose >250 mg/dL. Patients with type 1 diabetes mellitus or insulin-dependent diabetes are also excluded. A1c measurements are less reliable in leukemia patients due to anemia and/or need for red cell transfusions. Patients with well-controlled, non-insulin-dependent diabetes are eligible, but their blood glucose must be monitored closely during the study period in consultation with Diabetes specialists.
* Other severe acute, chronic medical, psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the treating physician, would make the patient inappropriate for entry into this study.
* Patients who cannot discontinue strong CYP3A inducers, grapefruit, grapefruit products, Seville oranges, or star fruit within the 3 days prior to starting venetoclax.

COHORT 2 Inclusion criteria

* Relapsed or refractory patients with acute leukemia with lymphoid lineage (B-ALL, T-ALL, ETP-ALL, mixed phenotype or bi-phenotypic) or lymphoblastic lymphoma (B- or T-lineage)

  * Bone marrow or peripheral blood involvement with ≥5% leukemic blasts. Patients with isolated extramedullary disease that is measurable by CT scan are also eligible.
* 18 years or older
* ECOG performance status 0-2
* Adequate organ function meeting protocol criteria
* Patients must be at least 2 weeks from major surgery or radiation therapy. A wash-out period of 5 half-lives is required for patients who participated in other investigational trials. These patients must have recovered from clinically significant toxicities related to these prior treatments.
* Patients must voluntarily sign and date an informed consent prior to the initiation of any screening or study-specific procedures.
* Females of childbearing potential will use effective contraception during protocol treatment and for at least 8 months after the last dose. Males with female partners of reproductive potential will use effective contraception during protocol treatment and for at least 5 months after the last dose.

Exclusion criteria

* Ph-positive ALL, Burkitt's leukemia/lymphoma
* Patient is pregnant or breastfeeding
* Patients with uncontrolled infection. Patients with infections that have been controlled for ≥7 days will be eligible.
* Known active hepatitis B or C infection, or uncontrolled human immunodeficiency virus (HIV) infection. Patients with HIV infection, whose disease is controlled with anti-retroviral therapy are eligible, but their highly active antiretroviral therapy (HAART) should be modified to minimize drug interactions. Due to the increased risk of hepatitis B reactivation, all patients with active, previously treated or resolved hepatitis B infection will not be eligible for rituximab treatment if their leukemia expresses >1% CD20.
* Major surgery or radiation therapy within 2 weeks prior to the first study dose
* Symptomatic central nervous system (CNS) disease or spinal cord compression
* Concurrent active malignancy requiring treatment with potential to influence the endpoint of the clinical trial. Patients with non-melanoma skin cancer, carcinoma in situ of the cervix, localized prostate cancer, past history of malignancy that has been definitively treated, and patients treated with hormonal therapies for solid tumors are eligible. Patients with history of multiple myeloma that does not need active treatment are also eligible.
* Uncontrolled cardiac disease
* Uncontrolled diabetes mellitus, defined as fasting blood glucose >160 mg/dL or random blood glucose >250 mg/dL. Patients with type 1 diabetes mellitus or insulin-dependent diabetes are also excluded. A1c measurements are less reliable in leukemia patients due to anemia and/or need for red cell transfusions. Patients with well-controlled, non-insulin-dependent diabetes are eligible, but their blood glucose must be monitored closely during the study period in consultation with Diabetes specialists.
* Other severe acute, chronic medical, psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the treating physician, would make the patient inappropriate for entry into this study.
* Patients who cannot discontinue strong CYP3A inducers, grapefruit, grapefruit products, Seville oranges, or star fruit within the 3 days prior to starting venetoclax.

Inclusion criteria

* Previously untreated patients with acute leukemia with lymphoid lineage (B-ALL, T-ALL, ETP-ALL, mixed phenotype or bi-phenotypic) or lymphoblastic lymphoma (B- or T-lineage)

  * Bone marrow or peripheral blood involvement with ≥20% leukemic blasts. Patients with isolated extramedullary disease that is measurable by CT scan are also eligible.
  * Previous therapy with dexamethasone or hydroxyurea given for cytoreductive purposes is allowed.
* 40 years old or older
* ECOG performance status 0-2
* Adequate organ function per protocol criteria
* Patients must be at least 2 weeks from major surgery.
* Patients must voluntarily sign and date an informed consent prior to the initiation of any screening or study-specific procedures.
* Females of childbearing potential will use effective contraception during protocol treatment and for at least 8 months after the last dose. Males with female partners of reproductive potential will use effective contraception during protocol treatment and for at least 5 months after the last dose.

Exclusion criteria

* Ph-positive ALL, Burkitt's leukemia/lymphoma
* Patient is pregnant or breastfeeding
* Patients with uncontrolled infection. Patients with infections that have been controlled for ≥7 days will be eligible.
* Known active hepatitis B or C infection, or uncontrolled human immunodeficiency virus (HIV) infection. Patients with HIV infection, whose disease is controlled with anti-retroviral therapy are eligible, but their highly active antiretroviral therapy (HAART) should be modified to minimize drug interactions. Due to the increased risk of hepatitis B reactivation, all patients with active, previously treated or resolved hepatitis B infection will not be eligible for rituximab treatment if their leukemia expresses >1% CD20.
* Major surgery or radiation therapy within 2 weeks prior to the first study dose
* Symptomatic central nervous system (CNS) disease or spinal cord compression
* Concurrent active malignancy requiring treatment with potential to influence the endpoint of the clinical trial. Patients with non-melanoma skin cancer, carcinoma in situ of the cervix, localized prostate cancer, past history of malignancy that has been definitively treated, and patients treated with hormonal therapies for solid tumors are eligible. Patients with history of multiple myeloma that does not need active treatment are also eligible.
* Uncontrolled cardiac disease
* Uncontrolled diabetes mellitus, defined as fasting blood glucose >160 mg/dL or random blood glucose >250 mg/dL. Patients with type 1 diabetes mellitus or insulin-dependent diabetes are also excluded. A1c measurements are less reliable in leukemia patients due to anemia and/or need for red cell transfusions. Patients with well-controlled, non-insulin-dependent diabetes are eligible, but their blood glucose must be monitored closely during the study period in consultation with Diabetes specialists.
* Other severe acute, chronic medical, psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the treating physician, would make the patient inappropriate for entry into this study.
* Any prior systemic chemotherapy or radiotherapy for treatment of ALL/LBL is an exclusion with the exception of hydroxyurea, steroids, ATRA and/or intrathecal chemotherapy. No more than 2 weeks of steroids is permitted.
* Patients who cannot discontinue strong CYP3A inducers, grapefruit, grapefruit products, Seville oranges, or star fruit within the 3 days prior to starting venetoclax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-03-17 (Estimated); Primary Completion 2032-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Safety of the combination of mini-hyperCVD and venetoclax plus capivasertib [Cohort 1] | After all cohort 1 participants have completed 2 28-day cycles of study treatment
  Summary of dose limiting toxicities as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Recommended Phase 2 Dose (RP2D) of capivasertib in combination with mini-hyperCVD and venetoclax [Cohort 1] | This will be assessed after all cohort 1 participants have completed 2 28-day cycles of study treatment
  The dose that dose not cause dose limiting toxicities as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5 will be identified as the RP2D.
Efficacy of capivasertib in combination with mini-hyperCVD and venetoclax [Cohort 2 and 3] | This will be assessed after all participants have completed treatment (an average of about 8 months)
  Number of participants with complete remission (CR) with measurable residual disease (MRD) negativity

SECONDARY OUTCOMES:
Rate of clinical remission (CR) [Cohort 1] | This will be assessed after all participants have completed treatment (an average of about 8 months)
Rate of clinical remission with incomplete count recovering (CRi) [Cohort 1] | This will be assessed after all participants have completed treatment (an average of about 8 months)
Rate of CR with measurable residual disease (MRD) negativity [Cohort 1] | This will be assessed after all participants have completed treatment (an average of about 8 months)
Progression free survival [All Cohorts] | up to 10 years after treatment completion
Overall survival [Cohort 2 and 3] | up to 10 years after treatment completion
Side effects of the combination of mini-hyperCVD and venetoclax plus capivasertib [Cohort 2 and 3] | This will be assessed after all participants have completed treatment (an average of about 8 months)
  Summary of dose limiting toxicities as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Caner Saygin, Study Chair — University of Chicago
Locations (1):
- University of Chicago Medicine Comprehensive Cancer Center, Chicago, Illinois, United States